CLINICAL TRIAL: NCT04688437
Title: Correlation Among Standing-sitting Sagittal Spinal Alignment, Paravertebral Muscle and Postoperative Clinical Outcomes in Patients With Adult Degenerative Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020322
Record Dates: First submitted 2020-12-18; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Degenerative Scoliosis
Keywords: Sitting; Standing; Sagittal alignment; Degenerative Scoliosis; Paravertebral Muscle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with degenerative scoliosis
  Interventions: Radiation: standard standing-sitting posteroanterior and lateral whole spine X-ray and lumbar MRI examination

INTERVENTIONS:
Radiation: standard standing-sitting posteroanterior and lateral whole spine X-ray and lumbar MRI examination — Routine examination

SUMMARY:
This is a prospective single-center study. Patients with adult degenerative scoliosis are prospectively enrolled and followed. All patients will take standard standing and sitting posteroanterior and lateral whole spine X-ray and lumbar MRI examination before and after surgery. Functional evaluation and radiographs were assessed preoperatively and postoperatively.This study will focus on the correlation among standing-sitting sagittal spinal alignment, paravertebral muscle and postoperative clinical outcomes in patients with adult degenerative scoliosis.

DETAILED DESCRIPTION:
The sagittal alignment of the spine, or sagittal balance, describe the ideal and normal sagittal spinal curvature distribution. With the deepening of the research on spinal morphology, function and pathology, more and more researchers pay attention to the role of sagittal alignment in the diagnosis and treatment of spinal deformity diseases. Some studies have shown that the restoration of patients with appropriate sagittal alignment can significantly improve their quality of life. Besides, paravertebral muscle can also influence the retaining of sagittal alignment. However, how to define the ideal sagittal alignment is still controversial for different patients with adult degenerative scoliosis(ADS) .

It was proved that the differences in sagittal parameters of the standing and sitting positions positions were influenced by age, gender and pelvic incidence(PI). In addition, patients with high PI are more prone to sagittal decompensation after long segment fixation (fixation of three or more segments) .Therefore, We speculate that the sagittal curvature of patients with large PI changes greatly from standing position to sitting position. So after long segment fixation, the spine in the state of standing position is more difficult to adapt to the changes of curvature and stress in sitting position, which is the possible reason that patients with high PI are more prone to sagittal decompensation. At present, how to design the proper corrective goals for patients according to both sagittal alignment and paravertebral muscle needs further research.

Thus, this study is aim to explore these three points about ADS patients: the characteristics of the sagittal spinal alignment changes from standing to sitting ; the adaption of the spine curvature in the standing and sitting position after long segment fixation surgery and the relationship among standing-sitting sagittal spinal alignment, paravertebral muscle and postoperative clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of adult degenerative scoliosis
* Cobb angle ≥10°

Exclusion Criteria:

* Neuromuscular diseases
* Arthritis
* Tumor
* A previous history of lumbar fusion surgery

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adult degenerative scoliosis who will undergo corrective surgery in Peking university third hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-20 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
The sagittal spinal parameters in degrees | 3 months after surgery
  The parameters included TPA (T1 pelvic angle,the angle between the line from the axis of the femoral head to the center of T1 and the line from the axis of the femoral head to the midpoint of the S1 endplate), lumbar lordosis (LL,the angle between the upper endplate of L1 and S1), thoracic kyphosis (TK,The angle between the upper endplate of T4 and the lower endplate of T12), pelvic incidence (PI,The angle between the line perpendicular to the midpoint of the sacral plate and the line connecting this to the midpoint of the hip axis), pelvic tilt (PT,The angle between the line from the middle of the sacral plate to the middle of the hip axis and the vertical line), sacral slope (SS,The angle between the sacral endplate and the horizontal line) Cobb angle of the curves
The sagittal spinal parameters in degrees | 6 months after surgery
  The parameters included TPA (T1 pelvic angle,the angle between the line from the axis of the femoral head to the center of T1 and the line from the axis of the femoral head to the midpoint of the S1 endplate), lumbar lordosis (LL,the angle between the upper endplate of L1 and S1), thoracic kyphosis (TK,The angle between the upper endplate of T4 and the lower endplate of T12), pelvic incidence (PI,The angle between the line perpendicular to the midpoint of the sacral plate and the line connecting this to the midpoint of the hip axis), pelvic tilt (PT,The angle between the line from the middle of the sacral plate to the middle of the hip axis and the vertical line), sacral slope (SS,The angle between the sacral endplate and the horizontal line) Cobb angle of the curves
The sagittal spinal parameters in degrees | 12 months after surgery
  The parameters included TPA (T1 pelvic angle,the angle between the line from the axis of the femoral head to the center of T1 and the line from the axis of the femoral head to the midpoint of the S1 endplate), lumbar lordosis (LL,the angle between the upper endplate of L1 and S1), thoracic kyphosis (TK,The angle between the upper endplate of T4 and the lower endplate of T12), pelvic incidence (PI,The angle between the line perpendicular to the midpoint of the sacral plate and the line connecting this to the midpoint of the hip axis), pelvic tilt (PT,The angle between the line from the middle of the sacral plate to the middle of the hip axis and the vertical line), sacral slope (SS,The angle between the sacral endplate and the horizontal line) Cobb angle of the curves
The sagittal spinal parameters in millimeters | 3 months after surgery
  SVA (sagittal vertical axis, The offset between the center of C7 and the plumb line drawn from posterosuperior corner of S1)
The sagittal spinal parameters in millimeters | 6 months after surgery
  SVA (sagittal vertical axis, The offset between the center of C7 and the plumb line drawn from posterosuperior corner of S1)
The sagittal spinal parameters in millimeters | 12 months after surgery
  SVA (sagittal vertical axis, The offset between the center of C7 and the plumb line drawn from posterosuperior corner of S1)
parameters of paraspinal muscles | 12 months after surgery
  the cross-sectional area (square centimeter)
parameters of paraspinal muscles | 12 months after surgery
  fatty infiltration rate of paraspinal muscles
functional outcomes of paraspinal muscles | 3 months after surgery
  the time of paraspinal muscle strength test
functional outcomes of paraspinal muscles | 6 months after surgery
  the time of paraspinal muscle strength test
functional outcomes of paraspinal muscles | 12 months after surgery
  the time of paraspinal muscle strength test

SECONDARY OUTCOMES:
Disability assessed by the Oswestry Disability Index (ODI) | 3 months after surgery; 6 months after surgery; 12 months after surgery;
  The Oswestry Disability Index (ODI) (0-100) is used to assess disability.Higher scores mean a worse outcome.
Disability assessed by the Japanese Orthopaedic Association (JOA) | 3 months after surgery; 6 months after surgery; 12 months after surgery;
  Japanese Orthopaedic Association (JOA)(-6-29) Scores is used to assess disability.Higher scores mean a better outcome.
Back pain assessed by the VAS | 3 months after surgery; 6 months after surgery; 12 months after surgery;
  The Visual Analog Scale (0-10) is used to evaluate back pain.Higher scores mean a worse outcome.
Leg pain assessed by the VAS | 3 months after surgery; 6 months after surgery; 12 months after surgery;
  The Visual Analog Scale (0-10) is used to evaluate leg pain.Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi Li, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lafage R, Schwab F, Challier V, Henry JK, Gum J, Smith J, Hostin R, Shaffrey C, Kim HJ, Ames C, Scheer J, Klineberg E, Bess S, Burton D, Lafage V; International Spine Study Group. Defining Spino-Pelvic Alignment Thresholds: Should Operative Goals in Adult Spinal Deformity Surgery Account for Age? Spine (Phila Pa 1976). 2016 Jan;41(1):62-8. doi: 10.1097/BRS.0000000000001171. PMID 26689395
- [Background] Zhou S, Xu F, Wang W, Zou D, Sun Z, Li W. Age-based normal sagittal alignment in Chinese asymptomatic adults: establishment of the relationships between pelvic incidence and other parameters. Eur Spine J. 2020 Mar;29(3):396-404. doi: 10.1007/s00586-019-06178-9. Epub 2019 Oct 29. PMID 31664567
- [Background] Hey HWD, Teo AQA, Tan KA, Ng LWN, Lau LL, Liu KG, Wong HK. How the spine differs in standing and in sitting-important considerations for correction of spinal deformity. Spine J. 2017 Jun;17(6):799-806. doi: 10.1016/j.spinee.2016.03.056. Epub 2016 Apr 7. PMID 27063999
- [Background] Zhou S, Sun Z, Li W, Wang W, Su T, Du C, Li W. The standing and sitting sagittal spinopelvic alignment of Chinese young and elderly population: does age influence the differences between the two positions? Eur Spine J. 2020 Mar;29(3):405-412. doi: 10.1007/s00586-019-06185-w. Epub 2019 Oct 19. PMID 31630266
- [Background] Cho KJ, Suk SI, Park SR, Kim JH, Kang SB, Kim HS, Oh SJ. Risk factors of sagittal decompensation after long posterior instrumentation and fusion for degenerative lumbar scoliosis. Spine (Phila Pa 1976). 2010 Aug 1;35(17):1595-601. doi: 10.1097/BRS.0b013e3181bdad89. PMID 20386505